CLINICAL TRIAL: NCT04459052
Title: Phase II: Physiological Effects of Nutritional Support in Patients With Parkinson's Disease
Brief Title: FDOPA PET and Nutritional Support in Parkinson's Disease
Acronym: FdopaPD2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: 20D.408
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Parkinson Disease; Idiopathic Parkinson Disease
Keywords: Alternative Medicine; Complementary Medicine; Parkinson's disease; Neurodegenerative Diseases; Idiopathic Parkinson's disease; Central Nervous System Diseases; Movement Disorders; N acetyl cysteine; [F-18] Fluorodopa; magnetic resonance spectroscopy; PET; positron emission tomography; dopaminergic function
MeSH Terms: conditions — Parkinson Disease; Neurodegenerative Diseases; Central Nervous System Diseases; Movement Disorders | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: This is an Open Label study. Randomization will occur via a 1:1 ratio of the NAC group and the waitlist control groups using the method of random permuted blocks with random block sizes without stratification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oral and IV N acetyl Cysteine Cohort (Other): Administration of Intravenous (IV) and Oral N-acetyl Cysteine (NAC) Intervention: IV NAC infusion: Dose: 50mg in 200ml of Dextrose 5% in Water (D5W), frequency: over one hour 1 x per week for 90 days ± 30 days AND Oral N-acetyl Cysteine - one 500 mg tablet 2 x per day (on days IV N-acetyl cysteine is not administered). Oral NAC will be taken for approximately 6 ±3 months.
  Interventions: Dietary Supplement: N acetyl cysteine; Drug: [F-18] Fluorodopa Positron Emission Tomography
- Waitlist Control Cohort (Other): Standard of Care Treatment for approximately 6 ±3 months.
  Interventions: Drug: [F-18] Fluorodopa Positron Emission Tomography

INTERVENTIONS:
Dietary Supplement: N acetyl cysteine — Intervention: IV NAC infusion: Dose: 50mg in 200ml of Dextrose 5% in Water (D5W), frequency: over one hour 1 x per week for 90 days ± 30 days AND Oral N-acetyl Cysteine - one 500 mg tablet 2 x per day (on days IV N-acetyl cysteine is not administered)
  Other Names: NAC
  Arms: Oral and IV N acetyl Cysteine Cohort
Drug: [F-18] Fluorodopa Positron Emission Tomography — FDOPA PET diagnostic imaging to to measure dopamine function, serum measures of NAC concentrations, magnetic resonance spectroscopy (MRS) to measure inflammatory and oxidative stress markers, and neurological measures to assess clinical symptoms, in patients with PD who are given oral capsules plus IV infusions of NAC in addition to standard of care for PD for 6 months.
  Other Names: FDOPA PET/MRI

SUMMARY:
The overall goal of this study will be to further our understanding of how N Acetyl Cysteine (NAC) can help to support dopaminergic function in patients with Parkinson's disease (PD). We plan to use pre and post Positron emission tomography magnetic resonance imaging (PET-MRI) with [F-18] Fluorodopa (FDOPA) to measure dopamine function, and neurological measures to assess clinical symptoms, in patients with PD who are given oral capsules plus IV infusions of NAC in addition to standard of care for PD for 6 ±3 months in an open label cross over design. Serum measures of NAC concentrations, magnetic resonance spectroscopy (MRS) to measure inflammatory and oxidative stress markers, may be conducted.

DETAILED DESCRIPTION:
The study consists of two arms in this crossover design study. The first arm of this study will receive intravenous and oral NAC, which is a strong antioxidant that increases brain glutathione, which may be beneficial in PD. NAC, is the N-acetyl derivative of the naturally occurring amino acid, L-cysteine. It is a common over-the-counter supplement and also is available as an injectable pharmaceutical that protects the liver in cases of acetaminophen overdose. Laboratory studies have displayed some benefits to use of NAC, such as its potential to counteract intracellular damage that leads to dopaminergic neuron death. It also has the potential to reduce markers of oxidative damage, protect against dopamine cell death from 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine (MPTP) toxicity, and to increase glutathione in blood, which might be useful in preventing oxidative damage in PD patients. The second arm will be a waitlist control receiving standard PD care. It should be noted that both arms will receive standard of care treatment for PD which will be augmented with NAC. A key component of this study is to evaluate the effects of NAC on dopamine, using PET imaging with FDOPA. Specifically, we will plan to study changes in dopamine levels before and after receiving approximately nutritional support with NAC.. This will allow us to evaluate whether NAC helps to support dopamine function. FDOPA PET imaging will be conducted at baseline and then after the nutritional support or standard of care for the waitlist arm. Then the waitlist group will receive NAC and the arm that received NAC initially will be crossed over to a standard of care group. FDOPA imaging will be conducted at the end of that period.

For evaluation of the dopamine function, [F-18] Fluorodopa (FDOPA), dose (5-10 millicurie (mCi), ± 20%) will be injected intravenously into an antecubital vein. Subjects will be premedicated with 200 mg of carbidopa orally approximately one hour prior to injection.

FDOPA has been available for over 30 years but has not been previously approved for commercial use by the FDA.We will be obtaining the FDOPA from the University of Pennsylvania cyclotron that has produced FDOPA for many Investigational New Drug applications (INDs) It will also be beneficial to assess whether there are specific changes in levels of different molecules that are related to energy consumption and oxidative stress. Proton MR spectroscopy (1H-MRS) has been previously performed in Parkinson's disease (PD) and parkinsonian syndromes to evaluate in vivo concentrations of basal ganglia and cerebral cortex metabolites such as N-acetylaspartate (NAA), choline (Cho), and creatine (Cr). We plan to include MRS as an additional biomarker to evaluate the potential effects of the nutritional supplements and/or NAC on oxidative stress and cerebral activity in PD patients.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of PD
2. Age 30 years old and older
3. Physically independent, ambulatory
4. Hoehn and Yahr score of I-III inclusive.
5. On stable antiparkinsonian medication for at least one month
6. Women of childbearing potential will confirm a negative pregnancy test and must practice effective contraception during the period of pilot study. In addition, male subjects who have a partner of childbearing age should practice effective contraception.

Exclusion Criteria:

1. Known allergy to NAC
2. Previous brain surgery.
3. Cognitive impairment by evaluation or known score on Mini-Mental Status examination of 25 or lower.
4. Wheelchair-bound or bed-ridden, non-ambulatory.
5. Intracranial abnormalities that may complicate interpretation of the brain scans (e.g., stroke, tumor, vascular abnormality affecting the target area).
6. History of head trauma with loss of consciousness > 48 hours.
7. Any medical disorder or physical condition that could reasonably be expected to interfere with the assessment of parkinsonian syndrome symptoms, or with any of the study assessments including the PET-MRI imaging.
8. Metal in the body that would prevent MRI scanning (as determined by the PI)
9. Patients with evidence of a significant psychiatric disorder by history/examination that would prevent completion of the study will not be allowed to participate.
10. Patients with current alcohol or drug abuse
11. Pregnant or lactating women.
12. Enrollment in active clinical trial/ experimental therapy within the prior 30 days.
13. Pending surgery during the course of the study.
14. History of thrombocytopenia or clotting disorders.
15. Cancer patients receiving active chemotherapy.
16. Severe gastroesophageal reflux disease.
17. History of uncontrolled diabetes, , gastroesophageal reflux disease, thyroid conditions
18. History of uncontrolled asthma.
19. History of severe kidney disease (if a patient reports this problem, a serum creatinine will be checked to assess glomerular filtration rate (GFR) and if it is less than 30, they will be excluded),
20. Patients taking medications that might interact with NAC involved in this study will be evaluated on a case-by-case basis by the PI or study physician. These medications include: Medications for high blood pressure; Medications that slow blood clotting; Medications for diabetes; Nitroglycerin.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-04-30 (Actual); Primary Completion 2025-04-11 (Actual); Study Completion 2027-01-08 (Estimated)

PRIMARY OUTCOMES:
FDOPA PET | Change from Baseline at approximately 6 months ± 3 months to access changes in Dopaminergic Function.
  To evaluate if intravenous/oral NAC helps to support dopamine function in the brain of
  patients with PD by using FDOPA PET imaging and subsequently helps to improve symptoms. Imaging will be conducted for standard of care and NAC arms.
FDOPA PET | Change from Baseline at approximately 12 months ± 3 months months to access changes in Dopaminergic Function.
  To evaluate if intravenous/oral NAC helps to support dopamine function in the brain of
  patients with PD by using FDOPA PET imaging and subsequently helps to improve symptoms. Imaging will be conducted for standard of care and NAC arms.

SECONDARY OUTCOMES:
Magnetic Resonance Spectroscopy (MRS) | Change from Baseline at approximately 6 months ± 3 months to access changes in oxidative stress and metabolism..
  To evaluate whether intravenous/oral NAC helps to support changes in oxidative stress and metabolism, as measured by magnetic resonance spectroscopy (MRS), in patients with PD in the standard of care and NAC arms of the study.
Magnetic Resonance Spectroscopy (MRS) | Change from Baseline at approximately 12 months ± 3 months to access changes in oxidative stress and metabolism..
  To evaluate whether intravenous/oral NAC helps to support changes in oxidative stress and metabolism, as measured by magnetic resonance spectroscopy (MRS), in patients with PD in the NAC and standard of care arms of the study.

OTHER OUTCOMES:
Blood Draw | .Change from Baseline NAC at approximately 6 months ± 3 months to assess serum concentration analysis of NAC.
  Blood draw may be conducted to perform a serum concentration analysis of NAC to confirm the levels of NAC achieved. The samples are obtained before and after receiving the first and last dose of NAC.
Unified Parkinson's Disease Rating Scale or Movement Disorders Scale | Change from Baseline at approximately 6 months ± 3 months to access changes in PD symptoms.
  Standardized assessment with the Unified Parkinson's Disease Rating Scale or Movement Disorders Scale to determine improvements in PD symptoms. A score of 199 on the UPDRS scale represents the worst symptoms with a score of zero representing no disability.
Unified Parkinson's Disease Rating Scale or Movement Disorders Scale | Change from Baseline at approximately 12 months to access changes in PD symptoms.
  Standardized assessment with the Unified Parkinson's Disease Rating Scale or Movement Disorders Scale to determine improvements in PD symptoms. A score of 199 on the UPDRS scale represents the worst symptoms, with a score of zero representing no disability.
Profile of Mood States | Change from Baseline at approximately 6 months ± 3 months to access changes anxiety and mood in PD symptoms.
  Profile of Mood States is a standardized self-report inventory will be administered to evaluate changes in mood, current state or traits. is a psychological rating scale used to assess transient, distinct mood states. The questionnaire contains 65 words that are rated on a scale of zero for not at all to 4 for extremely. There are 5 mood subscales: tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. A higher score for the total mood indicates a greater degree of mood disturbance.
Profile of Mood States | Change from Baseline at approximately 12 months ± 3 months to access changes anxiety and mood in PD symptoms.
  Profile of Mood States is a standardized self-report inventory will be administered to evaluate changes in mood, current state or traits. is a psychological rating scale used to assess transient, distinct mood states. The questionnaire contains 65 words that are rated on a scale of zero for not at all to 4 for extremely. There are 5 mood subscales: tension-anxiety, depression, anger-hostility, vigor, fatigue, and confusion. A higher score for the total mood indicates a greater degree of mood disturbance.
Beck Depression Inventory | Change from Baseline at approximately 6 months ± 3 months to access depression and changes in mood in PD symptoms.
  Beck Depression Inventory is a 21 question self report inventory to access depression and changes in mood. The highest possible total for the whole test would be 63; the lowest possible score for the test would be zero. A higher score indicates worse symptoms of depression and mood.
Beck Depression Inventory | Change from Baseline at approximately 12 months ± 3 months to access depression and changes in mood in PD symptoms.
  Beck Depression Inventory is a 21 question self report inventory to access depression and changes in mood. The highest possible total for the whole test would be 63; the lowest possible score for the test would be zero. A higher score indicates worse symptoms of depression and mood.
Parkinson's Disease Questionnaire-39. | approximately 6 months ± 3 months
  Parkinson's Disease Questionnaire-39 (PDQ).is a self report inventory that will be used to access changes in Parkinson's Disease symptoms. The total score for the PDQ is the sum of the scores for the 20 items. The highest possible total for the whole test would be 100; the lowest possible score for the test would be zero. Individual subscale scores for attention/concentration, retrospective memory, prospective memory, and planning/organization can also be generated by calculating the sum of specific sets of items. The highest possible total for the whole test would be 100; the lowest possible score for the test would be zero.
Parkinson's Disease Questionnaire-39. | approximately 12 months ± 3 months
  Parkinson's Disease Questionnaire-39 (PDQ).is a self report inventory that will be used to access changes in Parkinson's Disease symptoms. The total score for the PDQ is the sum of the scores for the 20 items. The highest possible total for the whole test would be 100; the lowest possible score for the test would be zero. Individual subscale scores for attention/concentration, retrospective memory, prospective memory, and planning/organization can also be generated by calculating the sum of specific sets of items. The highest possible total for the whole test would be 100; the lowest possible score for the test would be zero.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel A Monti, MD, MBA, Study Chair — TJU, Dept. Chair: Integrative Medicine and Nutritional Sciences
Locations (1):
- Thomas Jefferson University, Marcus Institute of Integrative Health Centers, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
After each participant completes the study, study scan data will be shared with co-investigators; participants may receive a copy of each scan after study completion.
Supporting Information: CSR
Time Frame: Study scan report will be offered to the subject after subject completes study
Access Criteria: Access only to authorized research staff and study participants

REFERENCES:
- [Background] Monti DA, Zabrecky G, Kremens D, Liang TW, Wintering NA, Cai J, Wei X, Bazzan AJ, Zhong L, Bowen B, Intenzo CM, Iacovitti L, Newberg AB. N-Acetyl Cysteine May Support Dopamine Neurons in Parkinson's Disease: Preliminary Clinical and Cell Line Data. PLoS One. 2016 Jun 16;11(6):e0157602. doi: 10.1371/journal.pone.0157602. eCollection 2016. PMID 27309537